CLINICAL TRIAL: NCT00288132
Title: Bridging Barriers to Diabetes Care With Telemedicine: The Diabetes TeleCare Study (DTC)
Brief Title: The Diabetes TeleCare Study
Acronym: DTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R18 67312 (completed); R18DK067312 (NIH)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; self-management; telemedicine; retinal; screening
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care
- Intervention (Experimental)
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — A 12-month diabetes self-management intervention delivered via telemedicine, with opportunity to receive telemedicine-based screening eye exam, was conducted.
  Arms: Intervention
Behavioral: Usual Care — Upon randomization, received one 15-minute diabetes self-management individual session, using American Diabetes Association materials. Continued care, as usual, from their primary care provider throughout duration of active 12 month intervention period.
  Arms: Usual Care

SUMMARY:
The American Diabetes Association clinical care guidelines stress the importance of metabolic control to prevent complications and improve quality of life for persons with diabetes. Unfortunately, these guidelines have not had widespread acceptance into clinical practice. Therefore, we propose translational research to evaluate telemedicine technology using interactive video conferencing (Diabetes TeleCare) as a novel means to increase the availability of health professionals in rural communities for the effective delivery of a diabetes self-management education program and as a means to provide retinal screenings in the primary care setting.

DETAILED DESCRIPTION:
According to recent 2002 estimates, the yearly cost of diabetes was approximately $132 billion. The burden of diabetes is considerable, particularly for ethnically diverse populations. Disease management programs that focus on self-management education have been effective in improving metabolic control. Accordingly, the American Diabetes Association clinical care guidelines stress the importance of metabolic control to prevent complications and improve quality of life for persons with this disease. Unfortunately, these advances have not resulted in widespread acceptance into clinical practice. Therefore, we propose translational research to evaluate telemedicine technology using interactive video conferencing (Diabetes TeleCare) as a novel means to increase the availability of health professionals in rural communities for the effective delivery of a diabetes self-management education program and as a means to provide retinal screenings in the primary care setting. Our aims are to 1) develop and implement a 12-month intervention, Diabetes TeleCare to improve adherence to diabetes clinical care guidelines and improve diabetes control in two community health centers located in ethnically diverse, rural and medically underserved communities, 2) conduct a one-year randomized clinical trial (RCT) of 200 patients to formally evaluate the effectiveness of Diabetes TeleCare compared to Usual Care in a sample with >60% African-Americans, and 3) determine the cost-effectiveness and satisfaction of Diabetes TeleCare compared to Usual Care. Participants are recruited from two community health centers in rural South Carolina and randomized according to a patient randomization schedule. Diabetes TeleCare (a structured curriculum) is delivered by a team consisting of a registered nurse/certified diabetes educator (RN-CDE) and an experienced registered dietitian, with support by other health professionals who are linked by interactive video conferencing to participants (single and group) in rural health centers at distant locations. The primary outcomes are measures of metabolic control (A1c, lipids), blood pressure, and use of the telemedicine-facilitated retinal screening capacity. Secondary outcomes include satisfaction, quality of life, health beliefs, and knowledge. The economic analysis will include an assessment of resource utilization, cost, and health utilities. In addition, incremental reductions in costs per A1c and the estimated lifetime cost-utility of Diabetes TeleCare compared to usual care will be determined. Telemedicine may be an effective alternative to traditional health care delivery systems resulting in improved diabetes education and control.

The intervention goal was to achieve an A1c <7%, with secondary goals of 10% weight loss and increasing exercise to at least 30 minutes a day, 5 days a week. Participants attend 13 sessions, 2 in the first month (1 group, 1 individual), monthly thereafter (9 group, 2 individual). Three group sessions were conducted in-person, all others were conducted via telemedicine. The self-management education team consisted of an RN/CDE and an RD. Sessions were conducted remotely, with a trained facilitator (LPN) at the clinic site. Participants were given a notebook and new material was added at each session. Completion of self-monitoring logs, including blood sugar, diet and physical activity, was assigned daily followed by less frequently based on progress towards intervention goals.

ELIGIBILITY:
Inclusion Criteria:

* All participants must have a confirmed physician diagnosis of type 2 diabetes supported by American Diabetes Association diagnostic criteria for blood glucose levels or
* Current use of oral hypoglycemic agents or insulin as confirmed by brief medical record review.
* All adults (> 21 years of age) who have a A1c value > 7.0 will be eligible.

Exclusion Criteria:

* Exclusion criteria applies to individuals with limitations that could limit safe participation in the study,

  * such as metastatic cancer,
  * multiple or recent (within six months) myocardial infarction (MI) or stroke,
  * dialysis for end stage renal disease,
  * severe psychiatric disease or dementia, or
  * inability to walk without an assistive device.
* We will also exclude women who are pregnant at the time of study recruitment (based on self report only) because of the unique needs related to diabetes self-management during pregnancy.
* We will, however, retain women in the study should they become pregnant during the course of the project.
* Individuals will be excluded if they plan to move out of the area.
* Additional exclusions may include inability to complete baseline tasks to the satisfaction of the lead interventionist or other more subjective assessment suggesting inability or unwillingness to adhere reasonably to the intervention based on interventionist review.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 6 mths, 12 mths, 24 mths

SECONDARY OUTCOMES:
Blood pressure | 6 mths, 12 mths, 24 mths
LDL Cholesterol | 6 mths, 12 mths, 24 mths
Cost effectiveness and cost utility | 6 mths, 12 mths
Retinal examination rates | 12 months
Weight | 6 mths, 12 mths, 24 mths
Waist Circumference | 6 mths, 12 mths, 24 mths

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Davis, MD, Principal Investigator — University of South Carolina
Locations (1):
- CareSouth Bennettsville, Bennettsville, South Carolina, United States

REFERENCES:
- [Result] Davis RM, Hitch AD, Salaam MM, Herman WH, Zimmer-Galler IE, Mayer-Davis EJ. TeleHealth improves diabetes self-management in an underserved community: diabetes TeleCare. Diabetes Care. 2010 Aug;33(8):1712-7. doi: 10.2337/dc09-1919. Epub 2010 May 18. PMID 20484125